CLINICAL TRIAL: NCT03402503
Title: A Randomized Phase IIa, Multi-center, Double-blind, Placebo-controlled Study to Assess the Safety, Feasibility, Tolerability, and Efficacy of a New Buccal Film of Montelukast in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Safety, and Efficacy of a New Buccal Film of Montelukast in Patients With Mild to Moderate Alzheimer's Disease
Acronym: BUENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IntelGenx Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IGX-CLI-2017-001
Record Dates: First submitted 2018-01-10; First posted 2018-01-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Montelukast buccal film, administered 10-mg once or 30-mg twice daily (once in the morning and once in the evening) for 26 weeks.
  Interventions: Drug: Montelukast buccal film
- Group B (Placebo Comparator): Placebo buccal film, administered once or twice daily (once in the morning and once in the evening) for 26 weeks.
  Interventions: Other: Placebo buccal film

INTERVENTIONS:
Drug: Montelukast buccal film — Film with active investigational product (montelukast) inserted and applied on inner cheek
  Arms: Group A
Other: Placebo buccal film — Film with placebo (no active drug) inserted and applied on inner cheek
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate the safety, feasibility, tolerability and efficacy of a new buccal film of montelukast in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized Phase IIa, multi-center, double-blind, placebo-controlled study of a new buccal film of montelukast in patients with mild to moderate Alzheimer's Disease. Study drug (montelukast or matching placebo) will be administered once or twice daily for 26 weeks, and treatment effect will be assessed primarily using the global NTB composite score at Week 26.

Patients who consent to participate will undergo screening assessments to determine eligibility. This study will enroll patients who are ≥50 years of age with mild to moderate Alzheimer's Disease and on a stable treatment of donepezil, rivastigmine or galantamine for ≥3 months. Patients will be randomized (using a balanced block randomization schedule) to one of two treatment groups:

* Group A: Montelukast buccal film
* Group B: Matching placebo buccal film

In addition to the global NTB composite, patients will also be evaluated using the MMSE, ADCS-CGIC, ADCS-ADL23, NPI and S-STS. Patients will be followed for any safety concerns throughout the study and for 4 weeks following the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate Alzheimer's Disease.
* MMSE score of 14 - 22
* CT or MRI within 18 months prior to screening indicating clinical phenotype of Alzheimer's Disease
* Treated daily with donepezil, rivastigmine or galantamine for ≥ 3 months
* All other medications for chronic conditions should have been at a stable dose for at least 2 weeks prior to first dose.
* No clinically meaningful abnormalities on electrocardiogram (ECG), physical examination and clinical laboratory tests

Exclusion Criteria:

* Taken memantine within 2 months prior to screening.
* Current diagnosis of any psychiatric disorder, depression that is not well-controlled, clinically significant or unstable systemic disease, or severe medical procedures
* Clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation.
* Patients at imminent risk of self-harm, based on clinical interview and response on S-STS
* History of malignancy occurring within 5 years immediately prior to screening, except for a subject who has been adequately treated for (1) basal cell or squamous cell skin cancer, (2) in situ cervical cancer, (3) localized prostate carcinoma, or (4) who has undergone potentially curative therapy with no evidence of recurrence for more than 3 years post-therapy, and who is deemed at low risk for recurrence by her/his treating physician
* History of any of the following cardiovascular conditions that an unstable:

  * Hypotension
  * Hypertension
  * Active cardiovascular disease
* Evidence of cerebrovascular disease
* Have used or plan to use the following medications from 30 days prior to Visit 1 through the end of the study:

  * Narcotic analgesics more frequently than on three days per week as needed for pain;
  * Daily antipsychotic (except for risperidone, quetiapine and aripiprazole, and only if at a stable and controlled dose)
  * Daily anxiolytic use; however, occasional use as needed for acute agitation or to be used as a rescue anxiolytic (i.e., lorazepam and oxazepam) is acceptable as long as not used within 24 hours of a clinic visit window;
  * Daily antidepressants (except for citalopram, escitalopram, venlafaxine, trazodone, sertraline, and mirtazapine, and only if at a stable and controlled dose);
  * Low potency antipsychotic agents (eg chlorpromazine) - not permitted at any time during the study;
  * Anti-parkinson's disease medications (selegiline, levodopa, amantadine) for the treatment of Parkinson's Syndrome Complex;
  * Lithium;
  * Clozapine;
* Previously treated with or currently using montelukast

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-04-03 (Actual)

PRIMARY OUTCOMES:
Global Neuropsychological test battery (NTB) Composite | To be conducted at Visit 2 (Baseline), Visit 4 (Week 6), Visit 6 (Week 12) and Visit 8 (Week 26)
  Evaluate if treatment with montelukast new buccal film is superior to placebo, assessed at Week 26 using the global NTB composite score. The NTB score will be used to assess cognitive and behavioral functions including problem-solving and conceptualization. The composite score will be based on an equally weighted average of standardized change from baseline scores on the following tests: International Shopping List Test (ISLT), ISLT-Delay, One Back Test, One Card Learning Test, Verbal Fluency Test, Category Fluency Test, Identification Test and Detection Test.

SECONDARY OUTCOMES:
Global Neuropsychological test battery (NTB) Composite | To be conducted at Visit 4 (Week 6) and Visit 6 (Week 12)
  Evaluate whether 6 and 12 weeks treatment with montelukast is superior to placebo, assessed using the global NTB composite scores. The NTB score will be used to assess cognitive and behavioral functions including problem-solving and conceptualization. he composite score will be based on an equally weighted average of standardized change from baseline scores on the following tests: International Shopping List Test (ISLT), ISLT-Delay, One Back Test, One Card Learning Test, Verbal Fluency Test, Category Fluency Test, Identification Test and Detection Test
Mini Mental State Examination (MMSE) | To be conducted at Visit 1 (Screening), Visit 2 (Baseline), Visit 4 (Week 6), Visit 6 (Week 12), Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast improved scores using the MMSE. The MMSE will be used to assess the subject's mental status in terms of cognitive function and level of dementia. The MMSE test will consist of an 11-question measure that will test five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30.
Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC) | To be conducted at Visit 2 (Baseline) and Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast improved scores using the ADCS-CGIC. ADCS-CGIC assessment and rating will be based on investigator's observation of changes in the subject's cognitive, functional, and behavioral performance since the beginning of a clinical trial (baseline) until end of treatment (Week 8).
Alzheimer's Disease Cooperative Study - Activities of Daily Living, 23-items scale (ADCS-ADL23) | To be conducted at Visit 2 (Baseline) and Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast improved scores using the ADCS-ADL23. The ADCS-ADL23 outcome measurement along with the assistance of the caregiver, will measure and evaluate the change from baseline and at Week 8, in the competence and performance of the subject in conducting their basic tasks and instrumental activities of daily living.
Neuropsychiatric Inventory (NPI) | To be conducted at Visit 2 (Baseline) and Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast improves the behavioral disturbance in patients, measured by the neuropsychiatric inventory (NPI), compared to placebo. NPI is an assessment of the frequency and severity of behavioral disturbances in dementia. The inventory comprises 10 behavioural areas: delusions, hallucinations, agitation/aggression, depression, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behaviour; and 2 neurovegetative areas. Each area has a screening question between 7 and 9 follow-up questions relating to symptoms, asked if the answer to the screening question was 'yes'. Ratings will be based on frequency, severity and distress on identified behaviours. The change from Baseline and at 26 week treatment will be measured.
Sheehan Suicide Tracking Scale (S-STS) | To be conducted at all visits i.e., Visit 1 (Screening), Visit 2 (Baseline), Visit 3 (Week 3), Visit 4 (Week 6),Visit 5 (Week 9), Visit 6 (Week 12), Visit 7 (Week 18), and Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast affected suicidal risk, measured by the S-STS.
Incontinency Frequency Rating | If there is a known history of incontinence, ratings to be conducted at all visits i.e., Visit 1 (Screening), Visit 2 (Baseline), Visit 3 (Week 3), Visit 4 (Week 6),Visit 5 (Week 9), Visit 6 (Week 12), Visit 7 (Week 18), and Visit 8 (Week 26)
  Evaluate whether 26 weeks of treatment with montelukast improved bladder incontinence in patients who reported this problem, measured by recording events and observations in the incontinency frequency rating.
Incidence of Treatment-Emergent Adverse Events | 26 Weeks
  Clinical safety and tolerability of montelukast film will be assessed up to Week 26 by adverse event monitoring (as assessed by CTCAE v5.0).

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Pietrantonio, PhD, Study Director — IntelGenx Corp.
Locations (12):
- Canada (12):
  - Vancouver Island Health Authority, Victoria, British Columbia
  - Centricity Research (formerly True North Clinical Research), Halifax, Nova Scotia
  - Centricity Research (formerly True North Clinical Research), New Minas, Nova Scotia
  - Bruyère Research Institute, Ottawa, Ontario
  - Recherches Neuro-Hippocampe, Ottawa, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - Gerontion Research Inc., Toronto, Ontario
  - Baycrest, Toronto, Ontario
  - Recherche Neuro-Hippocampe, Gatineau, Quebec
  - Centre hospitalier universitaire de Québec -Université Laval, Québec, Quebec
  - Centre de recherche sur le vieillissement, CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Undecided